CLINICAL TRIAL: NCT06546046
Title: Analysis of the Efficacy and Stability of a Single-Channel Patch-Type Wearable Electrocardiogram Monitor
Brief Title: Analysis of the Efficacy and Stability of a Wearable ECG Monitor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mezoo Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDV-2024-01
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Arrhythmias, Cardiac; Bradycardia; Tachycardia; Atrial Fibrillation; Atrial Flutter; Ventricular Premature Complexes
Keywords: Monitoring; Telemetry; Wearable device; Arrhythmia alarm; Signal loss; Satisfaction survey
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Tachycardia; Atrial Fibrillation; Atrial Flutter; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECG monitoring by telemetry device and patch-type ECG monitor at the same time (Experimental): The patient undergoes electrocardiogram monitoring simultaneously through a telemetry device and a patch-type electrocardiograph.
  Interventions: Device: ECG monitoring by telemetry device and patch-type ECG monitor at the same time

INTERVENTIONS:
Device: ECG monitoring by telemetry device and patch-type ECG monitor at the same time — The patient undergoes electrocardiogram monitoring simultaneously through a telemetry device and a patch-type electrocardiograph.

SUMMARY:
This study aims to analyze the efficacy and safety of wearable electrocardiogram (ECG) monitoring by simultaneously attaching a single-channel patch-type wearable ECG monitoring device (HiCardi+ by Mezoo Co., Ltd.) and a telemetry device (IntelliVue MX40 by Philips) used in actual wards to patients prescribed with ECG monitoring

DETAILED DESCRIPTION:
This study aims to analyze the efficacy and safety of wearable electrocardiogram (ECG) monitoring by simultaneously attaching a single-channel patch-type wearable ECG monitoring device (HiCardi+ by Mezoo Co., Ltd.) and a telemetry device (IntelliVue MX40 by Philips) used in actual wards to patients prescribed with ECG monitoring. After the data collection is completed, a satisfaction survey will be conducted with the medical staff. The data obtained simultaneously from HiCardi+ and MX40 will be analyzed, and the satisfaction survey responses from the medical staff will be reviewed to confirm the clinical convenience of the patch-type ECG monitoring device.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Patients admitted to Chonnam National University Hospital who require ECG monitoring
3. Individuals who have expressed their intention to participate in this study or have obtained written consent from a proxy

Exclusion Criteria:

1. Individuals who are unable to provide consent themselves or through a legally designated representative
2. Individuals deemed unsuitable for participation in the clinical trial based on the researcher's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The number of total QRS complex | Within 3 months after electrocardiogram monitoring procedure
  Number of total QRS complex is compared based on the data obtained simultaneously from two devices.
The rate of signal loss | Within 3 months after electrocardiogram monitoring procedure
  Rate of signal loss is compared based on the data obtained simultaneously from two devices.

SECONDARY OUTCOMES:
Average heart rate | Within 3 months after electrocardiogram monitoring procedure
  Average heart rate is compared based on the data obtained simultaneously from two devices.
The number of arrhythmia and technical alarm | Within 3 months after electrocardiogram monitoring procedure
  Number of arrhythmia and technical alarm is compared based on the data obtained simultaneously from two devices.
Results of satisfaction survey | Within 3 months after electrocardiogram monitoring procedure
  Satisfaction survey responses from the medical staff

REFERENCES:
- [Background] Choi W, Kim SH, Lee W, Kang SH, Yoon CH, Youn TJ, Chae IH. Comparison of Continuous ECG Monitoring by Wearable Patch Device and Conventional Telemonitoring Device. J Korean Med Sci. 2020 Nov 16;35(44):e363. doi: 10.3346/jkms.2020.35.e363. PMID 33200590
- [Background] Kwon S, Choi EK, Lee SR, Oh S, Song HS, Lee YS, Han SJ, Lim HE. Comparison of Novel Telemonitoring System Using the Single-lead Electrocardiogram Patch With Conventional Telemetry System. Korean Circ J. 2024 Mar;54(3):140-153. doi: 10.4070/kcj.2023.0252. PMID 38506104
- [Background] Marouf M, Vukomanovic G, Saranovac L, Bozic M. Multi-purpose ECG telemetry system. Biomed Eng Online. 2017 Jun 19;16(1):80. doi: 10.1186/s12938-017-0371-6. PMID 28629374
- [Background] Nelson BW, Allen NB. Accuracy of Consumer Wearable Heart Rate Measurement During an Ecologically Valid 24-Hour Period: Intraindividual Validation Study. JMIR Mhealth Uhealth. 2019 Mar 11;7(3):e10828. doi: 10.2196/10828. PMID 30855232